CLINICAL TRIAL: NCT05303844
Title: A Phase 1b Dose-escalation and Cohort-expansion Study of the Safety/Tolerability, and Efficacy of Oncolytic Virotherapy Plus PD-1 Inhibitor for Patients With Refractory Malignant Ascites (OPTIONS-02)
Brief Title: Oncolytic Virotherapy Plus PD-1 Inhibitor for Patients With Refractory Malignant Ascites
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Peng Wang, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2201249-7
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Refractory Malignant Ascites
MeSH Terms: interventions — tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- H101 + Tislelizumab (Experimental): (Dose escalation and cohort expansion) H101 administered by Intraperitoneal injection in combination with Tislelizumab administered intravenously (IV).
  Interventions: Drug: H101; Drug: Tislelizumab

INTERVENTIONS:
Drug: H101 — H101 intratumorally injection starts at day 0.
Drug: Tislelizumab — Tislelizumab will be initiated on day 1. Tislelizumab will be administered at 200 mg i.v. every 3 weeks until documented disease progression, development of unacceptable toxicity, participant request, or withdrawal of consent.

SUMMARY:
The objective of this study is to evaluate the safety/tolerability efficacy of oncolytic virotherapy combined with Tislelizumab for patients with refractory malignant ascites.

DETAILED DESCRIPTION:
This study is to evaluate the safety, effectiveness of local immune activation, and efficiency in patients with refractory malignant ascites after Intraperitoneal injection of oncolytic Viruses H101 and Tislelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained.
* Age ≥ 18 years at time of study entry.
* Pathologically diagnosed solid tumor malignancy.
* Malignant peritoneal ascites confirmed by peritoneal brush cytology.
* Failures from chemotherapy against malignant ascites.
* Cooperative Oncology Group-Status (ECOG Status) 0 or 1

Exclusion Criteria:

* Previous (<4 weeks) or concurrent treatment with systemic or intraperitoneal chemotherapy or biological agents such as monoclonal antibodies.
* History of cardiac disease, including clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment
* Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
* Prior treatment with oncolytic virotherapy.
* Radiotherapy administered less then 4 weeks prior to study treatment start.
* Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
* Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
* Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
* Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
* Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:
* history of interstitial lung disease
* Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
* known acute or chronic pancreatitis
* active tuberculosis
* any other active infection (viral, fungal or bacterial) requiring systemic therapy
* history of allogeneic tissue/solid organ transplant
* diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of Tislelizumab treatment.
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
* Live vaccine within 30 days prior to the first dose of Tislelizumab treatment or during study treatment.
* History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of Tislelizumab treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS
* Medication that is known to interfere with any of the agents applied in the trial.
* Any other efficacious cancer treatment except protocol specified treatment at study start.
* Patient has received any other investigational product within 28 days of study entry.
* Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.

Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-04-02 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Number of patient with dose-limiting toxicities (DLTs) as evaluated accordingly to CTCAE 5.0 | 28 days
  The DLT assessment period is defined as: Day of Injection through 28 days post injection (Safety Follow Up). A DLT will be defined as any Grade 3 or higher adverse event, as assessed by the National Cancer Institute Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.
Maximum tolerated dose (MTD) of intratumoral injection of H101 on at three dose levels in combination with anti-PD1 antibody. | 28 days
  A MTD is determined if any cohort experiences 2 subjects with DLT's.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | max 24 months

SECONDARY OUTCOMES:
Ascites Objective Response Rate | max 24 months
  The ascites objective response rate (ORR) was calculated as a summed ratio of patients with disappeared and decreased ascites to the total number of patients.
Objective Response Rate (ORR) | max 24 months
  ORR according to RECIST 1.1
Duration of Response | max 24 months
Progression Free Survival | max 24 months
Overall survival | max 42 months
disease control rate | max 24 months
Change from baseline local immune effects after H101 intraperitoneal injections | max 24 months
  Detection of increased local immune activation in malignant ascites will be assessed by single cell sequencing and/or Mass Cytometry (CyTOF).

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China